CLINICAL TRIAL: NCT04283565
Title: Health-economic Evaluation of the Care Pathway in General Medicine for High Cardiovascular Risk Patients Based on the Detection of Asymptomatic Lower Limb Peripherial Arterial Disease (AOMI) by the Blood Pressure Index (BPI).
Brief Title: Cost-utility Analysis, Cost-effectiveness Analysis, Budget Impact Analysis
Acronym: DAMAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: Collèges Régionaux de Médecine Générale- CRMG - 42270 ST PRIEST EN JAREZ (Unknown); Collèges Régionaux de Médecine Générale- CRMG - 26330 Châteauneuf-de-Galaure (Unknown); Collèges Régionaux de Médecine Générale- CRMG - 29238 BREST (Unknown); Collèges Régionaux de Médecine Générale- CRMG - 37400 Amboise (Unknown); Collèges Régionaux de Médecine Générale- CRMG - 59110 LA MADELEINE (Unknown); Collèges Régionaux de Médecine Générale- CRMG - 63 001 CLERMONT FERRAND (Unknown); Collèges Régionaux de Médecine Générale- CRMG - 18600 SANCOINS (Unknown); Collèges Régionaux de Médecine Générale- CRMG - 35000 Rennes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: PRM16-ER-DAMAGE
Record Dates: First submitted 2019-06-11; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Peripheral Arterial Disease
Keywords: detection; cost-utility analysis; cost-effectiveness analysis; blood pressure index measurement; motivational interviewing
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Two strategies are studied in this study:
  * Screening for asymptomatic AOMI by measuring IPS
  * Management of the FRCV by advices and motivational interviewing
  The strategies will be associated according to a factorial plan 2 * 2 in order to obtain 4 groups:
  * Strategy 1: Routine testing for asymptomatic AOMI and management of FRCV.
  * Strategy 2: Routine practice of asymptomatic AOMI screening and management of FRCVs by councils and a MA.
  * Strategy 3: Systematic Screening of asymptomatic AOMI by measurement of SPI and routine management of FRCV.
  * Strategy 4: Systematic screening of asymptomatic AOMI by measuring SPI and taking care of FRCVs by councils and a ME.
Masking Description: The investigators will include the patients before knowing their randomization arm. This procedure is essential to avoid selection bias by having an effect on the level of recruitment and the profile of the people included in the study.
  The initial randomization unit is the CRMG. Eight CRMG will be included in the investigator's study. Four CRMGs will be randomly assigned to the group "systematic AOMI screening by IPS measurement", four CRMG to the "no systematic screening" group. Then, each group thus obtained will be randomly divided into two CRMGs with "advice and EM" and two without CRMG.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Strategy 1: Usual practice (No Intervention): No systematic screening of asymptomatic AOMI and routine management of FRCV.
- Strategy 2: Motivationnal interviewing (Experimental): No systematic screening of asymptomatic AOMI and management of CVRF by a motivationnal interviewing.
  Interventions: Other: Management of CVRF by a motivationnal interviewing.
- Strategy 3: Systematic screening of AOMI by BPI measurement (Experimental): Systematic screening of AOMI by BPI measurement and routine management of FRCV.
  Interventions: Other: Systematic screening of AOMI by BPI measurement.
- Strategy 4: Both strategies (Experimental): Systematic screening of AOMI by BPI measurement and management of CVRF by a motivationnal interviewing.
  Interventions: Other: Systematic screening of AOMI by BPI measurement.; Other: Management of CVRF by a motivationnal interviewing.

INTERVENTIONS:
Other: Systematic screening of AOMI by BPI measurement. — The strategies will be associated according to a 2*2 factorial design in order to obtain 4 arms
  Arms: Strategy 3: Systematic screening of AOMI by BPI measurement; Strategy 4: Both strategies
Other: Management of CVRF by a motivationnal interviewing. — The strategies will be associated according to a 2*2 factorial design in order to obtain 4 arms
  Arms: Strategy 2: Motivationnal interviewing; Strategy 4: Both strategies

SUMMARY:
Cardiovascular pathologies (CV), the second leading cause of death just behind tumors, are particularly frequent in France and strongly mobilize the resources of the healthcare system (ambulatory and health facility). The French High Authority for Health (HAS) has defined major cardio-vascular risk factors (CVRF): smoking, high blood pressure (hypertension), elevated total cholesterol (TC) or LDL, decreased HDL cholesterol, type II diabetes and age, and predisposing CVRF or discussed: obesity, sedentary lifestyle, menopause, elevation of triglycerides and genetic factors.

Lower-linb peripherial arterial disease (AOMI), even if asymptomatic, involves systemic atherial disease, responsible for mortality irrespective of the presence of CVRF. The prevalence of asymptomatic AOMI is 10 to 20% beyond 55 years old, and the associated mortality is 18 to 30% at 5 years.

Individual screening is achievable by well-conducted clinical evaluation and systematic measurement of the simple, non-invasive Blood Pressure Index (BPI) in all subjects at risk. A BPI<0.9 indicates an event risk close to that of the symptomatic patient. However, if this strategy is recommended by the HAS, it is not carried out systematically in current practice. Therapeutic means available for the management of an asymptomatic AOMI are the identification and support for controllable CVRF such as smoking and nutrition (diet and physical activity) in the context of secondary prevention of atherosclerosis. Thus, the generalization of a systematique screening strategy of AOMI, allowing faster handling of CVRF by advices and Motivational Interviewing (MI), could have a significant impact, both clinically and economically.

Patients could also benefit from this support in terms of quality of life both on the physiological dimension (effect of weight loss, correction of disorders of cardiac function, etc.), that on the psychic dimension (well-being of patients, management of disorders anxious). However, few studies have evaluated the benefit of such a strategy in terms of quality-adjusted life years (QALYs),none did it on a cost recovery basis. No such studies have been conducted in France.

The feasibility of this project is based on the success of a pilot study conducted in Centre-Val de Loire region (France) in 2013. It showed that the implementation of a strategy of systematic screening of the asymptomatic AOMI based on the measurement of the BPI in high cardiovascular risk patients is feasible in current practice by general practitioners, and could be more efficient than interventions performed in current practice.

ELIGIBILITY:
Inclusion Criteria:

* Man over 50 and under 80 or woman over 60 and under 90 with at least 2 CVRF including at least 1 major CVRF (Major CVRF: Active or stopped smoking for less than 3 years; Type II treated or not treated Diabetes; Other CVRF: Family history: myocardial infarction, sudden death <55 years (male first degree relative) or <65 years (female first degree relative) or Cerebrovascular Stroke (CVA) < 45 years old; Dyslipidemia: LDL-cholesterol> 1.6 g/L and / or HDL-cholesterol <0.4 g/L; HTA (≥ 140/90 mmHg) for at least 6 months, balanced or not)
* Ability to benefit of an Motivational interviewing and to complete a quality of life questionnaire (fluent in french)
* Social insured patient
* Informed consent

Exclusion Criteria:

* History of cardiovascular event (symptomatic AOMI, acute coronary syndrome, stroke, transient ischemic attack ...), therefore patient already in tertiary prevention
* Patient included in another interventional study

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
ICUR between different screening and management strategies of peripherial arterial disease and cardio-vascular risk factors. | 10 years
  Incremental Cost-Utility Ratio (ICUR): Cost per QALY gained at 10 years from the collective and health insurance viewpoint. The quality of life data needed to calculate QALYs will be obtained from the EQ-5D questionnaire and extrapolated to 10 years based on the risk of CV event (SCORE) and prescribed treatments. The costs will be collected by a CRF.

SECONDARY OUTCOMES:
ICER between different screening and management strategies of peripherial arterial disease and cardio-vascular risk factors. | 10 years
  Incremental Cost-Effectiveness Ratio (ICER): Cost per prevented cardio-vascular event at 10 years from the collective and health insurance viewpoint. CV events at 10 years will be compute from the SCORE calculation at 2 years. The cost will be collected by a CRF.
ICER between different screening and management strategies of peripherial arterial disease and cardio-vascular risk factors. | 2 years
  ICER: Cost per SCORE point less at 2 years from the collective and health insurance viewpoint. The cost will be collected by a CRF.
Budget impact (in €) at 5 years | 5 years
  Budget impact at 5 years from the collective and health insurance viewpoint of the dissemination of the most efficient strategy. The cost will be collected by a CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien BRUEL, Dr, Principal Investigator — CRMG SAINT ETIENNE; Clarisse DIBAO DINA, Dr, Principal Investigator — CRMG TOURS; Thierry FARGE, Pr, Principal Investigator — CRMG LYON; Sophie LALANDE, Dr, Principal Investigator — CRMG BREST; Michel CUNIN, Dr, Principal Investigator — CRMG LILLE; Philippe VORILHON, Dr, Principal Investigator — CRMG CLERMONT FERRAND; Delphine RUBÉ, Dr, Principal Investigator — CRMG NANTES; Emmanuel ALLORY,, Dr, Principal Investigator — CRMG RENNES; Florent CROUZET,, Dr, Principal Investigator — MG SAINT ETIENNE (42210 Montrond-les-Bains); Julien FAVIER, Dr, Principal Investigator — MG SAINT ETIENNE (42300 ROANNE); Bastien LAVAL, Dr, Principal Investigator — MG SAINT ETIENNE (42800 GENILAC); Julien PEYRARD, Dr, Principal Investigator — MG SAINT ETIENNE (43 120 MONISTROL/LOIRE; Jean Philippe MELIZAN, Dr, Principal Investigator — MG SAINT ETIENNE (42260 St Martin la sauveté); Catherine PLOTTON,, Dr, Principal Investigator — MG SAINT ETIENNE (42230 ROCHE LA MOLIERE); Romain LAMOTTE, Dr, Principal Investigator — MG SAINT ETIENNE (69590 SAINT SYMPHORIEN SUR COISE); Hervé BONNEFOND, Dr, Principal Investigator — MG SAINT ETIENNE (42000 SAINT ETIENNE); Alexandre BRULET, Dr, Principal Investigator — MG SAINT ETIENNE (42300 ROANNE); Olivier DURIEUX, Dr, Principal Investigator — MG SAINT ETIENNE (43240 SAINT JUST MALMONT); Claire CHARRAT, Dr, Principal Investigator — MG SAINT ETIENNE (43120 MONISTROL SUR LOIRE); Morinne DUPIN, Dr, Principal Investigator — MG SAINT ETIENNE (43210 BAS EN BASSET); Aurélien BARADEL, Dr, Principal Investigator — MG LYON (01430 ST MARTIN DU FRESNE); Myriam OLIVIA, Dr, Principal Investigator — MG LYON (38 280 VILLETTE D'ANTHON); Damien MONLOUBOU, Dr, Principal Investigator — MG LYON (69100 VILLEURBANNE); Ronan FOURE,, Dr, Principal Investigator — MG LYON (01160 PONT D'AIN); Nadia HASSAOUI,, Dr, Principal Investigator — MG LYON (01160 PONT D'AIN); Mélanie MICHEL, Dr, Principal Investigator — MG LYON (01160 PONT D'AIN); Pierre DE HAAS, Dr, Principal Investigator — MG LYON (01160 PONT D'AIN); Chloé FAYSSE, Dr, Principal Investigator — MG LYON (26750 CHATILLON ST JEAN); Christophe PIGACHE, Dr, Principal Investigator — MG LYON (26330 CHATEAUNEUF DE GALAURE); Gérard PETIT, Dr, Principal Investigator — MG LYON (69007 LYON); Emilie BECK ROBERT, Dr, Principal Investigator — MG BREST (29620 LANMEUR); Hélène CRENN CORVEZ, Dr, Principal Investigator — MG BREST (29620 LANMEUR); Etienne MELOT,, Dr, Principal Investigator — MG BREST (22420 LE VIEUX MARCHE); Lucas BEURTON- COURAUD,, Dr, Principal Investigator — MG BREST (29190 PLEYBEN); Aldric LUCAS, Dr, Principal Investigator — MG BREST (29190 PLEYBEN); Anton ROBIN YANN, Dr, Principal Investigator — MG BREST (29 000 QUIMPER); Pierre- Marie BOSSER, Dr, Principal Investigator — MG BREST (29790 PONT CROIX); Roberto PITMAN, Dr, Principal Investigator — MG BREST (29 400 LANDIVISIAU); Patrick BIARD, Dr, Principal Investigator — MG TOURS (37210 VOUVRAY); Julie GROSSE, Dr, Principal Investigator — MG TOURS (37400 AMBOISE); Aude LINASSIER, Dr, Principal Investigator — MG TOURS (37000 TOURS); Anne- Catherine SCHLEGEL, Dr, Principal Investigator — MG TOURS (37210 PARCAY MESLAY); Yann TEISSET, Dr, Principal Investigator — MG TOURS (37360 ROUZIERS DE TOURAINE); Sylvie TIERCIN, Dr, Principal Investigator — MG TOURS (37000 TOURS); Jean- Christophe TUROT, Dr, Principal Investigator — MG TOURS (37300 JOUE LES TOURS); Maxime PAUTRAT, Dr, Principal Investigator — MG TOURS (37240 LIGUEIL); Olivier CUVILLIER, Dr, Principal Investigator — MG TOURS (37390 LA MEMBROLLE SUR CHOISILLE); Ludivine BARBEAU, Dr, Principal Investigator — MG TOURS (41 7000 CHEVERNY); Anita TILLY, Dr, Principal Investigator — MG LILLE (59280 BOIS GRENIER); Ludovic WILLEMS, Dr, Principal Investigator — MG LILLE (59190 HAZEBROUCK); Laurent TURI, Dr, Principal Investigator — MG LILLE (62130 GAUCHIN VERLOINGT); Nassir MESSAADI, Dr, Principal Investigator — MG LILLE (59000 LILLE); Marc BAYEN, Dr, Principal Investigator — MG LILLE (59287 GUESNAIN); Axel DESCAMPS, Dr, Principal Investigator — MG LILLE (59770 MARLY); Sabine BAYEN, Dr, Principal Investigator — MG LILLE (59287 GUESNAIN); Jonathan FAVRE, Dr, Principal Investigator — MG LILLE (59650 VILLENEUVE D'ASCQ); Christian HULIN, Dr, Principal Investigator — MG LILLE (62000 ARRAS); Jan BARAN, Dr, Principal Investigator — MG LILLE (59150 WATTRELOS); Benoît CAMBON, Dr, Principal Investigator — MG CLERMONT FERRAND (03 800 GANNAT); Mathilde VICARD OLAGNE, Dr, Principal Investigator — MG CLERMONT FERRAND (63 580 LE VERNET LA NARENNE); Frédéric TESSIERES, Dr, Principal Investigator — MG CLERMONT FERRAND (43 100 BRIOUDE); Thibault MENINI, Dr, Principal Investigator — MG CLERMONT FERRAND (63 230 PONTGIBAUD); Yves NICOLLIN, Dr, Principal Investigator — MG CLERMONT FERRAND (63 500 ISSOIRE); Syndie CANN, Dr, Principal Investigator — MG BREST (29 520 CHATEAUNEUF DU FAVU); Gilles TANGUY, Dr, Principal Investigator — MG CLERMONT FERRAND (63 380 PONTAUMUR); Philippe MESTRE, Dr, Principal Investigator — MG CLERMONT FERRAND (43410 LEMPDES); PHILIPPE ZEGANADIN, Dr, Principal Investigator — MG CLERMONT FERRAND (63190 LEZOUX); Véronique BERTRAND JARROUSSE, Dr, Principal Investigator — MG CLERMONT FERRAND (6393 AUGEROLLES); Audrey MORICE RAMAT, Dr, Principal Investigator — MG NANTES (44118 LA CHEVROLIERE); Sylvain FOURE, Dr, Principal Investigator — MG NANTES (85000 LA ROCHE SUR YON); Chrystelle PEYRON, Dr, Principal Investigator — MG NANTES (44160 PONTCHATEAU); Mariette RABAUD PELLETIER, Dr, Principal Investigator — MG NANTES (85340 OLONNE SUR MER); Elodie COSSET, Dr, Principal Investigator — MG NANTES (85430 LES CLOUZEAUX); Brigitte TREGOUET, Dr, Principal Investigator — MG NANTES (85000 LA ROCHE SUR YON); Cécile RABILLER, Dr, Principal Investigator — MG NANTES (85430 LES CLOUZEAUX); Cédric RAT, Dr, Principal Investigator — MG NANTES (44000 NANTES); Antoine DE GUIBERT, Dr, Principal Investigator — MG RENNES (35000 RENNES); Mathilde GUERIN, Dr, Principal Investigator — MG RENNES (22690 PLEUDIHEN SUR RANCE); Isabelle EZANNO, Dr, Principal Investigator — MG RENNES (56950 CRACH); Gilles TAPIN, Dr, Principal Investigator — MG RENNES (35590 L'HERMITAGE); jean- François RICONO, Dr, Principal Investigator — MG RENNES (35560 ANTRAIN); Laure FIQUET, Dr, Principal Investigator — MG RENNES (35160 BRETEIL); Anne DONCIEUX, Dr, Principal Investigator — MG RENNES (56500 MOREAC); Hervé LE NEEL, Dr, Principal Investigator — MG RENNES (35200 RENNES); Stephane DUQUENNE, Dr, Principal Investigator — MG RENNES (56240 PLOUAY); Boris LAGOUTTE, Dr, Principal Investigator — 35250 ST AUBIN D'AUBIGNE